CLINICAL TRIAL: NCT06149104
Title: A Multicenter, Open-label Study to Collect the Safety Information of Sacubitril/Valsartan in Japanese Pediatric Patients With Heart Failure Due to Systemic Left Ventricle Systolic Dysfunction Who Have Completed CLCZ696B2319E1 Study
Brief Title: A Safety Study of Sacubitril/Valsartan in Japanese Pediatric Patients With Heart Failure Due to Systemic Left Ventricle Systolic Dysfunction Who Have Completed CLCZ696B2319E1 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696B2319E2
Record Dates: First submitted 2023-11-13; First posted 2023-11-28 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
Keywords: sacubitril/valsartan; post-trial access; pediatric; heart failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sacubitril/valsartan (Experimental): The starting dose of study drug was determined by the investigator in consideration of the participant´s condition. The dose level at the end of study visit of CLCZ696B2319E1 study could remain the same, or the dose level could be changed at the discretion of the investigator.
  Interventions: Drug: sacubitril/valsartan

INTERVENTIONS:
Drug: sacubitril/valsartan — sacubiril/valsartan

SUMMARY:
The purpose of this open-label study was to collect additional safety information of sacubitril/valsartan and to provide post-trial access to sacubitril/valsartan for the eligible Japanese patients who completed CLCZ696B2319E1(NCT03785405) study until marketed product of pediatric formulation, film-coated granules in capsule, is available in Japan.

DETAILED DESCRIPTION:
This trial (CLCZ696B2319E2) was a multicenter, open-label extension study for Japanese patients who have successfully completed the CLCZ696B2319E1 study. Only Japanese patients who successfully completed CLCZ696B2319E1 study and fulfilled protocol requirements were eligible to participate in this study.

The first visit (Visit Day1) was the same day as the End of Study visit of CLCZ696B2319E1 study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* <18 years of age (at the time of signing informed consent)
* Completed CLCZ696B2319E1 study and safely enrolled

Exclusion Criteria:

* Permanently discontinued the study treatment during CLCZ696B2319E1 study
* Renal vascular hypertension (including renal artery stenosis)
* History of angioedema
* Having parents or legal guardians who do not give consent or allow the child to give assent, or inability of patient or the parents/legal guardians to follow instructions or comply with follow-up procedures
* Any medical condition(s) that may put the patient at risk in the Investigator's opinion or that the Investigator deems unsuitable for the study

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Japan (6):
  - Novartis Investigative Site, Ōbu, Aichi-ken
  - Novartis Investigative Site, Ōmura, Nagasaki
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Toyama

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2538

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 6 investigative sites in Japan.
Pre-assignment Details: All consenting participants were assessed for eligibility into this study at the first visit (Visit Day 1) and the study medication was initiated.
Groups:
- Sacubitril/Valsartan: The starting dose of study drug was determined by the investigator in consideration of the participant´s condition. The dose level at the end of study visit of CLCZ696B2319E1 study could remain the same, or the dose level could be changed at the discretion of the investigator. All participants had a target dose of 3.1 mg/kg bid. If a participant was unable to tolerate up-titration to a higher sacubitril/valsartan dose level or at the discretion of the Investigator, participants could be maintained on lower dose levels of sacubitril/valsartan.
Period: Overall Study
Arm/Group | Sacubitril/Valsartan
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sacubitril/Valsartan
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.75 (4.234)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent adverse events (any AE regardless of seriousness), and SAEs.
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment, up to a maximum duration of approximately 8 months.
Population: Safety Set (SAF): all participants who received at least one dose of open-label study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sacubitril/Valsartan
Number analyzed (Participants) | 8
Participants
  Adverse Events | 6
  Serious Adverse Events | 1

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment, up to a maximum duration of approximately 8 months.
Groups:
- All Patients: All Patients
Arm/Group | Sacubitril/Valsartan | All Patients
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/8
Other Adverse Events (participants affected / at risk) | 6/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacubitril/Valsartan (N=8) | All Patients (N=8)
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacubitril/Valsartan (N=8) | All Patients (N=8)
Vomiting (Gastrointestinal disorders) | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 1
COVID-19 (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2
Otitis media (Infections and infestations) | 1 | 1
Streptococcal infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT06149104/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT06149104/SAP_001.pdf